CLINICAL TRIAL: NCT06716476
Title: Impact of Vitamin D in Modulating Disease Activity and Inflammatory Mediators in Rheumatoid Arthritis
Brief Title: Impact of Vitamin D in Rheumatoid Arthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pristina (Other)
Responsible Party: Principal Investigator, Shaip Krasniqi, Prof. Dr. Med. Shaip Krasniqi - Clinical Pharmacologist, University of Pristina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UPristina
Record Dates: First submitted 2024-11-22; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Rheumatic Arthritis
Keywords: Modulating Disease Activity and Inflammatory mediators
MeSH Terms: conditions — Rheumatic Fever | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment with Vitamin D (Active Comparator): RA Patients with Vitamin D
  Interventions: Drug: Vitamin D
- No treatment with Vitamin D (No Intervention): RA Patients without Vitamin D

INTERVENTIONS:
Drug: Vitamin D — Supplemental with Vitamin D 4000 IU
  Arms: Treatment with Vitamin D

SUMMARY:
The goal of this prospective, randomized, parallel-group design, double-blind, and 6-month follow-up is to evaluate the impact of 4000 IU/day vitamin D on 25-hydroxyvitamin D [25(OH)D] levels and inflammatory mediators in people with Rheumatoid Arthritis (RA).

The main questions it aims to answer are

* The level of 25(OH)D and inflammatory mediators of levels of RA differs at baseline and after 6 months of Vitamin D 4000 UI
* The disease activity of AR measured by visual analogue scale (VAS) and Disease Activity Score-28 (DAS-28 score) will change in baseline and after 6 months of Vitamin D 4000 UI Researchers will compare the group of participants with Vitamin D supplementation and group of participants without D Vitamin supplementation

Participants in active group will:

* Take Vitamin D every day for 6 months
* Visit the clinic in the first months and after 6 months for medical visits and tests.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is an idiopathic autoimmune disease with a chronic course of exacerbations and remissions with more frequent incidence in females, characterized by inflammation, pain, and progressive damage to the joints. The main focus of our study is to evaluate the impact of Vitamin D besides other standard therapies in the group of people with RA, assessing the inflammatory mediators and clinical course of the disease in the baseline and after six months.

This is a prospective, randomized, controlled Trial (RCT) with a Parallel-Group Design, ensuring that changes in inflammation markers and disease activity over time will be measured simultaneously and independently.

Before enrolment, the research dossier, including the patient's informed consent, was submitted to the Medical Chamber of Kosovo Ethics Committee for approval. This professional body approved this study, and the approval letter was issued to the research team. Patients were included in the study only after signing the consent form and after being fully informed about the research.

The participants will be patients which fulfils the diagnostic criteria for Rheumatoid Arthritis (RA) of American college of Rheumatology (ACR)/European league against rheumatism (EULAR) - ACR/EULAR 2010. The cohort of participants will be elected after evaluation of inclusion and exclusion criteria of participants:

The trial participants will be enrolled from a cohort of people with RA disease treated at the University Clinical Centre of Kosovo-Rheumatology Clinic in Prishtina. The data will be collected for one year.

In both group of participants at the baseline will be measured the level of 25-hydroxyvitamin D [25(OH)D] and inflammatory mediators of RA: Interleukin 6 (IL6) , Interleukin 17 (IL17), CRP, TNF-alpha). Moreover, in both groups participants will be determined the activity of disease measuring the visual analogue scale (VAS) and Disease Activity Score-28 (DAS-28 score). The intervention group of participants will receive the Vitamin D supplementation for 6 months while other group of participants will not receive the Vitamin D and after 6 months will be evaluated level of [25(OH)D] and inflammatory mediators of RA: Interleukin 6 (IL6) , Interleukin 17 (IL17), CRP, TNF-alpha) and VAS and Das28 and compare with baseline data.

ELIGIBILITY:
Inclusion criteria

* Rheumatoid Arthritis Caucasian patients,
* Kosovar ethnicity,
* Both genders,

Inclusion criteria:

* Patients with proven rheumatoid arthritis diagnosis ACR/EULAR 2010 grouped into four classifications with point scores for each:

  * joint symptoms;
  * serology (including RF and/or ACPA);
  * symptom duration, whether <6 weeks or >6 weeks; and
  * acute-phase reactants (CRP and/or ESR). Point scores ≥6/10 was criteria for AR diagnosis;
* RA disease duration 1-14 years

Exclusion criteria:

* Other inflammatory diseases;
* Thyroid and parathyroid diseases;
* Liver and kidney disease;
* Last 3 months treatment with Ca > 1g/per day;
* Last 3 months treatment with vitamin D supplements

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Level of 25(OH)D in serum | 6 months
  25(OH)D level in ng/mL (0-30 ng/mL)
Serum level of inflammatory mediators of RA (IL6, IL17, CRP, TNF-alpha) | 6 months
  IL-6 pg/mL < 12.0 IL-17 (pg/mL) <1.4 pg/mL TNF Alpha (pg/mL) 4.6 - 12.4 pg/mL CRP (mg/l) <6mg/L

SECONDARY OUTCOMES:
VAS: Visual analogue scale | 6 months
  The Visual Analogue Scale (VAS) measures pain intensity. The measurement unit 0 - 10 unit.
  The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be')
DAS28: Disease Activity Score-28 | 6 months
  The DAS28 is a measure of disease activity in RA; an online tool collates a clinical assessment of 28 specified joints, serum inflammatory markers, and a visual analog scale (0-10) of the patient's global function. A score greater than 5.1 indicates active disease and less than 3.2 indicates well-controlled disease.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine University of Prishtina, Pristina, Kosovo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Higgins MJ, Mackie SL, Thalayasingam N, Bingham SJ, Hamilton J, Kelly CA. The effect of vitamin D levels on the assessment of disease activity in rheumatoid arthritis. Clin Rheumatol. 2013 Jun;32(6):863-7. doi: 10.1007/s10067-013-2174-x. Epub 2013 Jan 23. PMID 23340834
- [Background] Chandrashekara S, Patted A. Role of vitamin D supplementation in improving disease activity in rheumatoid arthritis: An exploratory study. Int J Rheum Dis. 2017 Jul;20(7):825-831. doi: 10.1111/1756-185X.12770. Epub 2015 Oct 20. PMID 26481198
- [Background] Fassio A, Gatti D, Rossini M, Bertelle D, Bixio R, Viapiana O, Milleri S, Benini C, Pistillo F, Zanetti G, Adami G. Effects on Serum Inflammatory Cytokines of Cholecalciferol Supplementation in Healthy Subjects with Vitamin D Deficiency. Nutrients. 2022 Nov 14;14(22):4823. doi: 10.3390/nu14224823. PMID 36432510
- [Background] Adams JS, Hewison M. Unexpected actions of vitamin D: new perspectives on the regulation of innate and adaptive immunity. Nat Clin Pract Endocrinol Metab. 2008 Feb;4(2):80-90. doi: 10.1038/ncpendmet0716. PMID 18212810
- [Background] Al-Saoodi H, Kolahdooz F, Andersen JR, Jalili M. Effect of vitamin D on inflammatory and clinical outcomes in patients with rheumatoid arthritis: a systematic review and dose-response meta-analysis of randomized controlled trials. Nutr Rev. 2024 Apr 12;82(5):600-611. doi: 10.1093/nutrit/nuad083. PMID 37437898
- [Background] Steiner G, Van Hoovels L, Csige D, Gatto M, Iagnocco A, Szekanecz Z. Should ACR/EULAR criteria be revised changing the RF and ACPA scores? Autoimmun Rev. 2024 Jan;23(1):103421. doi: 10.1016/j.autrev.2023.103421. Epub 2023 Aug 24. PMID 37633353
- [Derived] Rexhepi M, Krasniqi B, Hoti K, Daci A, Rexhepi-Kelmendi B, Krasniqi S. Impact of vitamin D supplementation on disease activity and pain management in rheumatoid arthritis: a randomized double-blinded controlled study. BMC Rheumatol. 2025 Jul 11;9(1):87. doi: 10.1186/s41927-025-00543-6. PMID 40646666